CLINICAL TRIAL: NCT00327223
Title: A Phase 1 Trial of Amplimexon® (Imexon, Inj.) Administered Daily for 5 Days Every 3 Weeks to Patients With Metastatic Cancer or Disseminated Malignancy
Brief Title: Safety Study of Imexon Treatment of Patients With Metastatic or Disseminated Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AmpliMed Corporation (Industry)
Responsible Party: Evan Hersh, VP Medical Affairs, AmpliMed Corporation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP-011
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Neoplasm Metastasis
Keywords: Metastatic cancer; Disseminated malignant disease
MeSH Terms: conditions — Neoplasm Metastasis | interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imexon (Experimental): Dose escalation of imexon
  Interventions: Drug: imexon

INTERVENTIONS:
Drug: imexon

SUMMARY:
AMP-011 is a Phase 1 study designed to extend the understanding of the toxicity and pharmacology of imexon by investigating a schedule of daily treatment for 5 days every three weeks. The objective of the study is to determine the maximally tolerated dose, the pharmacokinetics, and the toxicity of the drug on the designated schedule.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated malignant disease of any type.
* Prior treatment; at least one prior regimen required.
* Able to perform the activities of daily living.
* Off prior cancer therapy for at least 4 weeks.
* If female, neither pregnant nor nursing.
* Willing to use contraceptives to prevent pregnancy.
* No other serious illnesses.
* No other active malignancy.
* No serious infections.
* No other current drug therapy for the cancer.
* Blood counts and blood chemistries in or near normal range.
* Prior radiation is permitted.

Exclusion Criteria:

* No active brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Determine the maximally tolerated dose
determine the pharmacokinetics
determine the toxicity of the drug on the designated schedule

CONTACTS AND LOCATIONS:
Overall Officials: Evan Hersh, MD, Study Director — AmpliMed Corporation
Locations (4):
- United States (4):
  - US Oncology Indiana, Indianapolis, Indiana
  - US Oncology Albany, New York Oncology, Albany, New York
  - Investigational Site 014, Temple, Texas
  - US Oncology, Tyler Cancer Center, Tyler, Texas